CLINICAL TRIAL: NCT03139409
Title: Digital Radiography in Detection of Recurrent Caries Underneath Chlorhexidine Containing Adhesive Versus Conventional Adhesive After One Year Follow up.
Brief Title: Digital Radiography in Detection of Recurrent Caries Underneath Chlorhexidine Containing Adhesive Versus Conventional Adhesive After One Year Follow up: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Katreen Tawfik, Internal Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-044-16
Record Dates: First submitted 2017-04-30; First posted 2017-05-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Caries Incidence
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventonal adhesive (Active Comparator): peak lc bond
  Interventions: Procedure: adhesive bond with chlorhexidine
- Time variable (Other): Diagnosis and follow up will be immediate ,6 months later and 1 year
  Interventions: Other: Time variable

INTERVENTIONS:
Procedure: adhesive bond with chlorhexidine — Peak® Universal Bond (ultradent, 505 West 10200 South, South Jordan, UT 84095،USA ) light-Cured Adhesive with Chlorhexidine (0.2%), 7.5% filler, phosphate and containing hydroxyethyl methacrylate with ethyl alcohol as the carrier. its viscosity has been optimized for minimal film thickness (2μm) and superior strength. using self etch adhesive with chlorexidine as one step in the bonding component may give chance to proper penetration of resin tags, decrease the micro-organisms due to the antibacterial effect of chlorexidine (Bin-Shuwaish, 2016) and also the addition of chlorexidine in bonding system may be an excellent tool to increase the stability of collagen fibrils within the hybrid layer against host-derived metaloproteinases (MMP) without the need for additional steps for the bonding protocol (Stanislawczuk, et al., 2009), which results in better durability and good restorations with decreasing the incidence of recurrent caries
  Other Names: peak universal bond
  Arms: conventonal adhesive
Other: Time variable — Diagnosis and follow up will be immediate , 6 months later and 1 year
  Arms: Time variable

SUMMARY:
This study will be conducted to compare the effect of chlorexidine containing adhesive versus conventional one in prevention of secondary caries lesion underneath composite restoration over one year follow up null hypothesis

DETAILED DESCRIPTION:
each patient will have at least 2 class II cavities.one will be restored using the intervention and the other using the control.

Digital radiographs will be taken and the images will be processed using a digital system. Then the teeth will be evaluated by expert in dental radiology who had no awareness of the results of the visual inspection. The examiner will use a radiograph viewer and a radiographic film magnifier to determine the presence or absence of radiolucency underlying the restoration. The clinical and radiographic examination will be assessed according to the FDI World Dental Federation clinical criteria for the evaluation of direct and indirect restorations The aim of this equivalent trial is to examine if the chlorhexidine containing adhesive is effective as the conventional adhesive in prevention of recurrent caries under resin composite restoration after one year follow up in high caries risk patients with class II cavities. Based on the previous papers by Papagiannoulis et al .,1999 and kohler et al.,2000, the success rate reported was about 95% (absence of caries). If there is truly no difference between the standard and experimental treatment, then 37 patients are required to be 80% sure that the limits of a two-sided 90% confidence interval will exclude a difference between the standard and experimental group of more than 15 %. The sample size was calculated by sealed envelope online.

Data will be analyzed using IBM SPSS advanced statistics (statistical package for social sciences), version 21 ( SPSS Inc. Chicago , IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Comparisons between categorical variables will be performed using the chi square test. An equivalent limit will be tested. A P -value less than or equal 0.05 will be considered statistically significant. All tests will be two tailed

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 20-25 years of age with high caries risk. Patients should have an acceptable oral hygiene level. Patients must have at least two proximal lesions to be restored.

Exclusion Criteria:

Patients with a compromised medical history. Severe or active periodontal disease. Heavy bruxism or a traumatic occlusion. Lack of compliance

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
recurrent caries incidence | 1 year
  FDI clinical and radiographic criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral Medicine and Dentistry, Cairo, Egypt